CLINICAL TRIAL: NCT00909064
Title: The Effects of Arixtra on Wound Drainage Following Total Joint Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Paul Di Cesare,MD (Other)
Responsible Party: Sponsor-Investigator, Paul Di Cesare,MD, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200816251; GSK576428
Record Dates: First submitted 2009-05-22; First posted 2009-05-27 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2009-05

CONDITIONS: Total Knee Replacement
MeSH Terms: interventions — Fondaparinux

ARMS (1):
- Arixtra (Experimental): Effect of Arixtra on would drainage and length of stay for the patients with hip and knee replacement
  Interventions: Drug: Fondaparinux Sodium (Arixtra)

INTERVENTIONS:
Drug: Fondaparinux Sodium (Arixtra) — 2.5 mg once per day to begin 6-8 hours after surgery and continued for 10 days.
  Other Names: Arixtra

SUMMARY:
The investigators hypothesize that Arixtra patients will be less likely to experience wound infection than patients who have received low-molecular weight heparin, coumadin or aspirin with mechanical compression.

ELIGIBILITY:
Inclusion Criteria:

* All primary unilateral TKA and THA cases will be included.

Exclusion Criteria:

* Patients less than 50 kg, Patients with CrCl<30ml/min. Revision and bilateral procedures will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul E. DiCesare, MD, Principal Investigator — University of California, Davis Health System
Locations (1):
- U C Davis, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arixtra
Started | 114
Completed | 114
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arixtra
Number analyzed (Participants) | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Days Until a Dry Wound
Description: Days from day of surgery to stoppage of leakage from the wound
Time Frame: Up to 10 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arixtra
Number analyzed (Participants) | 114
days | 3.6 (2.2)

2. Secondary Outcome: Number of Days in Hospital.
Description: Days after surgery to dischage
Time Frame: Up to 10 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arixtra
Number analyzed (Participants) | 114
days | 3.73 (1.4)

3. Secondary Outcome: Incidence of Wound Infection
Description: Incidence of Cellulitis in patients undergoing Arixtra treatment
Time Frame: Up to 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arixtra
Number analyzed (Participants) | 114
Participants | 2

ADVERSE EVENTS:
Time Frame: Length of hospital stay up to 10 days
Arm/Group | Arixtra
All-Cause Mortality (participants affected / at risk) | 0/114
Serious Adverse Events (participants affected / at risk) | 0/114
Other Adverse Events (participants affected / at risk) | 2/114
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arixtra (N=114)
Cellulitis (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes